CLINICAL TRIAL: NCT06721650
Title: Effect of Perturbation-Based Balance Training on Trunk Proprioception and Balance in Hemiplegic Cerebral Palsy: a Randomized Controlled Trial
Brief Title: Perturbation-Based Balance Training on Trunk Proprioception and Balance in Cerebral Palsy:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lama Saad El-Din Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Lama Saad El-Din Mahmoud, Assistant Professor of Neurology and Neurosurgery Faculty of Physical Therapy October 6 University, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005471
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Other)
  Interventions: Other: Perturbation-Based Balance Training; Other: the selected physical therapy exercise program
- control group (Other)
  Interventions: Other: the selected physical therapy exercise program

INTERVENTIONS:
Other: Perturbation-Based Balance Training — Perturbation-based balance training (PBT; or reactive balance training or perturbation training) is balance training that uses repeated, externally applied mechanical perturbations to trigger rapid reactions to regain postural stability in a safe and controlled environment
  Arms: study group
Other: the selected physical therapy exercise program — trunk control therapeutic exercise, static and dynamic balance treaining exercises

SUMMARY:
To investigate the effect of Perturbation-Based Balance Training on trunk proprioception and balance in hemiparetic cerebral palsy

DETAILED DESCRIPTION:
Thirty-eight patients with hemiplegic cerebral palsy will participate in this study.

The patients will randomly be divided into two equal groups; the control group which received the selected physical therapy exercise program and the study group received the same exercise training program in addition to Perturbation-Based Balance Training, three times per week for three months. The evaluation methods are BIODEX, The Pediatric Balance Scale, baseline digital inclinometer.

ELIGIBILITY:
Inclusion Criteria:

* - Thirty-eight children hemiplegic cerebral palsy
* Age will range as (8:10) years old
* Spastic hemiplegic cerebral palsy
* Normal body mass index ranged from 1SD to -2SDaccording to BMI-for age Z score charts include an age and sex- specific BMI for children (WHO, 2007).
* Gross motor function classification system: level I&II

Exclusion Criteria:

* • Difficulty to communicate or to understand program instructions

  * any other neurological deficits or orthopaedic abnormalities,
  * secondary musculoskeletal complication
  * vestibular problems
  * any mental impairment

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
BIODEX balance system | three months
  to evaluate postural balance. The BBS is a multiaxial device that objectively measures and records an individual's ability to stabilize the involved joint under dynamic stress.
Pediatric Balance Scale | three months
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points
baseline digital inclinometer. | four weeks
  for measuring lateral movement in applications like: Earth movement in the landslide zone. Detecting shear planes in hydraulic structures. Measuring stability during construction

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Giza, El-Sheikh Zayed City Giza 1133 Egypt, Egypt